CLINICAL TRIAL: NCT05000918
Title: Functional Food Application of Okara Protein Hydrolysate (OPH)- for Anti-exercise-fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Taichung University of Education (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CS2-20042
Record Dates: First submitted 2021-07-27; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPH group (Experimental): Participants should eat a pack of OPH once a day for 28 days. The dosage of the OPH is 11.74 g/day.
  Interventions: Dietary Supplement: Okara protein hydrolysate (OPH)

INTERVENTIONS:
Dietary Supplement: Okara protein hydrolysate (OPH) — Okara protein hydrolysate (OPH) was a pack of dried beige powder. It can be stored at room temperature, but it must be exposed to direct sunlight.

SUMMARY:
The aim of this study is to investigate the anti-exercise-fatigue effects of okara protein hydrolysate (OPH) in men

DETAILED DESCRIPTION:
Each subject must undergo a cardiopulmonary capacity test to assess the maximum oxygen uptake 1 week before the intervention (day 1), and then eat the test food for 4 weeks (day 8 to day 35). Before and after the intervention (the 8th and 35th day), posture measurement, diet questionnaire survey and endurance exercise ability test were carried out. The trial period was 35 days. The subjects will take blood samples before, during, after, and 30 minutes and 60 minutes after the end of the two endurance exercise tests. During the whole period of participating in the program, blood will be collected 10 times, each with a blood volume of 15 mL. Gas is collected during the period and within 1 hour after exercise. Gas is collected every 15 minutes and 1 minute at a time. Analyze his exercise time, oxygen intake and blood biochemical value.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male and aged 20-40.
* The subject has a usual exercise habit (exercising 2 times or more per week) and did not participate in professional sports competitions or professional sports training during the study period.
* No smoking or drinking habits.
* No food allergies and the liver function is normal.
* No cardiovascular diseases or other chronic diseases, and no serious illnesses requiring hospitalization during the study period.
* The subject can understand the test process described in the consent form and the possible potential risks and benefits, and can sign the consent form.
* The subject can accept dietary control during the trial period.

Exclusion Criteria:

* Those who have taken nutritional supplements containing branched-chain amino acids.
* Those who cannot complete the endurance exercise ability test.
* Those who are diagnosed with kidney disease, heart disease, or cancer and are still under active treatment.
* Have used other drugs, whose pharmacological effects may affect fatigue.
* Subjects who have systemic infections and require systemic antibiotics.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change the metabolic substances level after intervention | 8th day, 35th day
  Compare the difference of blood lactate, lactate dehydrogenase, and creatine kinase level after exercise between pre- and post-intervention

SECONDARY OUTCOMES:
Change the exercise time after intervention | 8th day, 35th day
  Compare the exercise time between pre- and post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan

IPD SHARING:
Plan to Share IPD: No